CLINICAL TRIAL: NCT01116674
Title: Pediatric Critical Illness Hyperglycemia and Glycemic Control Registry: A Project to Assist in the Improved Understanding of Hyperglycemia and Glycemic Control in Pediatric Critical Illness.
Brief Title: Pediatric Critical Illness Hyperglycemia and Glycemic Control Registry
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00045186; R21DK081847 (NIH); CIH Registry (Other: Other)
Record Dates: First submitted 2010-05-03; First posted 2010-05-05 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Hypoglycemia Hyperglycemia
Keywords: Intensive critical care, glycemic control, hypoglycemia, hyperglycemia , insulin treatment, intensive care outcomes, pediatrics
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Glycemic Control: Critically ill children at participating centers who require select vital organ support measure (i.e. mechanical ventilation, vasopressor, or continuous renal replacement therapy) will have routine blood glucose (BG) screening initiated (i.e. at least q 12 hours). If a patient has a BG reading of > 140 mg/dL, a repeat BG will be obtained in 1-2 hours. If this second BG is > 140 mg/dL the patient will be diagnosed with critical illness hyperglycemia and an insulin infusion will be started and BG will be maintained between 80-140 using a pediatric specific developed and tested algorithm.

SUMMARY:
The objective in this project is to assemble a consortium of pediatric critical care centers of varying size, acuity, and composition to evaluate our glycemic control protocol on at least 250 children with hyperglycemia in different critical care units.

***This Study is supported by an R21 Grant (MRR) from the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK).

DETAILED DESCRIPTION:
Many studies over the past decade have demonstrated that clinical outcomes can be improved in critically ill adults by aggressive management of hyperglycemic with insulin infusions (Van Den Berghe 2001, Van Den Berghe 2006, Krinsey 2004, Treggari 2008, Scalea, 2007, Lang 2007). Yet, in some of these studies and other recent trials (i.e. Glucontrol (Preiser, 2009) VISEP (Brunkhorst, 2008) and (NICE-SUGAR, 2009)), have highlighted the potential and real risks of glycemic control (namely iatrogenic hypoglycemia) and questioned how effectively glucose can be controlled in critical illness. One reason for the suboptimal glycemic control witnessed in some trials may be not rigorously refined and validated. Even as such, many medical oversight committees (including the Institutes of Healthcare Improvement, the American Diabetes Association, and Society of Critical Care Medicine, among others) continue to recommend regular and aggressive glycemic control in critically ill patients. Although not specifically included nor excluded from such recommendations, most pediatric intensivists have not incorporated glycemic control into regular practice primarily due to concerns of therapy induced hyperglycemia - although there are reports of protocols that appear to be effective at controlling BG levels with low rates of hypoglycemia (Preissig et al 2008, Verhoeven et al 2009).

Our group at Emory University and Children's' Healthcare of Atlanta has taken a progressive, yet methodical, approach to better understand the implications of hyperglycemia and its treatment in critically ill and injured children. Practitioners at our facility developed a pediatric-specific protocol to identify and treat hyperglycemia in critically ill children. We have instituted this approach as standard care in our facility and have experience with managing several hundred children with hyperglycemia. Our approach to glycemic management has very promising safety and efficacy profiles, even when compared to the most stringent and successful glycemic control protocols used in adults. We published the first experience in pediatric glycemic control in pediatric in 2008 (Preissig et al PCCM 2008) and have used our experience to identify specific risk factors for developing hypoglycemia (Preissig et al JPed, 2009).

The goal of this proposal is to assist our step-wise approach in investigating hyperglycemia in critically ill children by externally validating our glycemic control protocol via multi-center evaluation. In doing so, we will also be developing the infrastructure and a tested intervention that can be leveraged for future studies of hyperglycemia in pediatric critical illness, including a multi-center outcome trial. The specific hypothesis for this project is that our protocol is safe and efficient at identifying and managing hyperglycemia in critically ill or injured children in pediatric ICUs regardless of ICU size, acuity, model, staffing makeup, or clinical focus.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill children requiring mechanical ventilation, vasopressor/inotropes, continuous renal replacement therapy or other criteria, will have glycemic screening initiated. (Such are the risk factors that have been demonstrated to assist in the identification of critically children who will develop hyperglycemia (Preissig et al., JPeds., 2009)
* Admission to the pediatric medical/surgical or pediatric cardiac intensive care unit
* Require mechanical ventilation (endotracheal or via tracheotomy) and/or vasopressors/inotropic infusions (including dopamine, dobutamine, norepinephrine, epinephrine, vasopressin, or milrinone)
* Patient or family member available to discuss informed consent criteria and provide informed consent.

Exclusion Criteria:

* Patients with type I diabetes mellitus presenting to the ICU in diabetic ketoacidosis (DKA)
* Preexisting conditions in which there is impaired glycogen stores or counter regulatory response (i.e. inborn error of metabolism, fulminant hepatic failure)

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Childern upto 18 or 21 years old admitted to pedaitric intensive care units who are ar risk for deleveloping critical illness hyperglycemia.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Identify and manage hyperglycemia in pediatric intensive care unit | 5-2012
  Determine safety (ie hypoglycemia) and effectiveness (ie ability to establish/maintain glycemic control) of our pedatric-specific approach to control critical illness hyperglycemia.

SECONDARY OUTCOMES:
Consortium of centers practiced at glycemic control in pediatric intensive care unit. | 5-2012
  To develop a consortium of centers that will be practiced at glycemic control who may be able to participate in a future multi-center trial in glycemic control. To use the experience of other centers to refine a generalizable protocol to successfully and safely control hyperglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Rigby, MD, PhD, Principal Investigator — Emory University and Children's Healthcare of Atlanta at Egleston; Cathering M Preissig, MD (Co-I), Study Director — Medical Center of Central Georgia; Kevin O Maher, MD (Co-I), Study Director — Emory University and Children's Healthcare of Atlanta at Egleston; Daniel C Keeton, BA (Coordinator), Study Director — Children's Healthcare of Atlanta at Egleston and Emory University; Jeryl Huckaby, RRT (Coordinator), Study Director — Children's Healthcare of Atlanta at Egleston and Emory University
Locations (3):
- United States (3):
  - Children's Healthcare of Atlanta at Egleston - Pediatric Cardiac Intensive Care Unit, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Egleston - Pediatric Intensive Care Unit, Atlanta, Georgia
  - Medical Center of Central Georgia - Pediatric Intensive Care Unit, Macon, Georgia

REFERENCES:
- [Background] Preissig CM, Rigby MR, Maher KO. Glycemic control for postoperative pediatric cardiac patients. Pediatr Cardiol. 2009 Nov;30(8):1098-104. doi: 10.1007/s00246-009-9512-4. Epub 2009 Aug 25. PMID 19705188
- [Background] Preissig CM, Rigby MR. Pediatric critical illness hyperglycemia: risk factors associated with development and severity of hyperglycemia in critically ill children. J Pediatr. 2009 Nov;155(5):734-9. doi: 10.1016/j.jpeds.2009.05.007. Epub 2009 Jul 22. PMID 19628220
- [Background] Preissig CM, Rigby MR. A disparity between physician attitudes and practice regarding hyperglycemia in pediatric intensive care units in the United States: a survey on actual practice habits. Crit Care. 2010;14(1):R11. doi: 10.1186/cc8865. Epub 2010 Feb 3. PMID 20128893
- [Background] Preissig CM, Hansen I, Roerig PL, Rigby MR. A protocolized approach to identify and manage hyperglycemia in a pediatric critical care unit. Pediatr Crit Care Med. 2008 Nov;9(6):581-8. doi: 10.1097/PCC.0b013e31818d36cb. PMID 18838924